CLINICAL TRIAL: NCT06269224
Title: Examining Factors Influencing Thoracolumbar Mobility in Amateur Runners and Sedentary Individuals
Brief Title: Examining Factors Influencing Thoracolumbar Mobility in Runners
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Sarıoğlu, Principal Investigator, Hacettepe University
Other Study IDs: HU-FTR-KS-01
Record Dates: First submitted 2024-02-11; First posted 2024-02-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Runners; Mobility; Fascia; Range of Motion
Keywords: running; Latissimus Dorsi; Tone; Elasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- There are 3 groups. 2 groups consist of runners and 1 group consists of sedentary individuals.: Participants were recreational runners who run between 20 to 50 km weekly; one group consisted of 35 runners who had been RTY, the second group consisted of 35 runners who had been running for RSM; the third group was composed of 35 sedentary individuals identified using the Sedentary Behavior Questionnaire. Participants were within the age range of 30 to 45. Exclusion criteria encompassed a history of lower extremity or lumbar-related surgery within the last year and a body mass index (BMI) exceeding the normal threshold of 24.5 kg/m².
  Interventions: Other: Participants were recreational runners who run between 20 to 50 km weekly; each one has 35 runners.

INTERVENTIONS:
Other: Participants were recreational runners who run between 20 to 50 km weekly; each one has 35 runners. — The Myoton device was used over the Latissimus Dorsi (LD) muscle on both dominant and nondominant sides to measure muscle tone (Hz), elasticity, and stiffness (N/m) values. Trunk flexibility and flexibility of lumbar extensor muscles were measured with tape measurement (cm). The trunk range of motion (ROM, ˚) was measured using goniometer. Thoracolumbar Fascia Length Test and Modified Schober Test were used for thoracolumbar (TLF) fascia flexibility. The weekly training distance (km), duration (h) and daily water consumption (lt) rates were recorded. The percentage of individuals experiencing lower extremity injuries and lower back pain within the RSM group was calculated.

SUMMARY:
The presence of to is thoracolumbar (TL) mobility a significant aspect in the context of running. Most of the factors may be related to certain kinematic parameters of the lumbopelvic-hip complex during running.

DETAILED DESCRIPTION:
Context: The presence of to is thoracolumbar (TL) mobility a significant aspect in the context of running. Most of the factors may be related to certain kinematic parameters of the lumbopelvic-hip complex during running. Objective: To compare the TL mobility of individuals at different running levels and sedentary individuals. Design: Cross-sectional. Participants: The first group consisted of 35 runners who had been running for the last two years (RTY) while the second group had 35 runners who had been running for the last six months (RSM). The third group had 35 sedentary individuals. Main Outcomes Measures: Sports-related and sociodemographic information was recorded. The Myoton device was used over the Latissimus Dorsi (LD) muscle on both dominant and nondominant sides to measure muscle tone (Hz), elasticity, and stiffness (N/m) values. Trunk flexibility and flexibility of lumbar extensor muscles were measured with tape measurement (cm). The trunk range of motion (ROM, ˚) was measured using goniometer. Thoracolumbar Fascia Length Test and Modified Schober Test were used for thoracolumbar (TLF) fascia flexibility. Analysis of variance was used for statistical analysis. SPSS version 17.0 was used for all statistical analyses. The primary outcome was defined as lumbar extensor tightness. Numeric data obtained from the subjects were presented as mean, standard deviation (mean±SD) and percentage (%). The primary outcome was defined as lumbar extensor tightness. The sample size for each group was calculated to be 30 with a power of 80% and a significance level of 0.05. Considering potential dropouts, 35 participants were included in each group. The groups were not homogenous. As a nonparametric test, the 'Kruskal-Wallis test' was employed for the three-group comparison. The Mann-Whitney U test was used for the two-group comparison. Statistical significance was set at P < .05.

ELIGIBILITY:
Inclusion Criteria:

* The participants were within the age range of 30 to 45.

Exclusion Criteria:

* The history of lower extremity or lumbar-related surgery within the last year and a body mass index (BMI) exceeding the normal threshold of 24.5 kg/m².

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The participants were recreational runners who run between 20 to 50 km weekly. The first group consisted of 35 runners who had been running for the last two years (RTY) while the second group had 35 runners who had been running for the last six months (RSM).
  The third group was composed of 35 sedentary individuals identified using the Sedentary Behavior Questionnaire.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Myoton Assessment | 1 month
  The passive mechanical properties of the muscle (Tone, Stiffness, and Elasticity) were measured using the Myoton-3 myotonometer medical device (Myoton Ltd., Estonia, EU) (ICC: 0.80-0.93). The patients were positioned prone with a thin rolled towel placed under their foreheads and their arms in a 180˚ flexion position for a fifteen-minute period of rest. In our study, a point 5 cm below the lower tip of the scapula was identified along the imaginary line of the LD muscle. The probe was at a 90˚ angle to the skin. The measurements were repeated ten times at one-second intervals and the average values were recorded. These values were then calculated for dominant and nondominant sides.

CONTACTS AND LOCATIONS:
Overall Officials: Hacettepe University, Study Director — university
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't study for a doctorate. I want the data to remain private. But I will share my results. I think it will be enough to give my opinion in the discussion part.